CLINICAL TRIAL: NCT03432884
Title: A Two-Part Study Consisting of a Randomized, Placebo-Controlled, Single Dose Safety and Tolerability Study (Part A) Evaluating a Supratherapeutic Dose of Zanubrutinib Followed by a Randomized, Placebo- and Positive-Controlled, Crossover Study (Part B) to Evaluate the Effect of Zanubrutinib on Cardiac Repolarization in Healthy Volunteers
Brief Title: A Two-Part Phase 1 Study to Investigate the Safety and Tolerability of Supratherapeutic Dose of Zanubrutinib and Effect of Zanubrutinib on Cardiac Repolarization in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BGB-3111-106
Record Dates: First submitted 2018-01-19; First posted 2018-02-14 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; pharmacokinetics; safety
MeSH Terms: interventions — zanubrutinib; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Part A: Single Group Part B: Crossover
Who Masked: Participant, Investigator
Masking Description: Part A: zanubrutinib and placebo will be double-blind Part B: zanubrutinib and placebo will be double-blind; Moxifloxacin will be open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: BGB-3111 (Experimental)
  Interventions: Drug: BGB-3111
- Part A: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B: BGB-3111, Placebo, and Moxifloxicin (Experimental)
  Interventions: Drug: BGB-3111; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: BGB-3111 — Subjects will receive BGB-3111
  Arms: Part A: BGB-3111; Part B: BGB-3111, Placebo, and Moxifloxicin
Drug: Placebo — Subjects will receive Placebo
  Arms: Part A: Placebo; Part B: BGB-3111, Placebo, and Moxifloxicin
Drug: Moxifloxacin — Subjects will receive Moxifloxicin
  Other Names: Avelox
  Arms: Part B: BGB-3111, Placebo, and Moxifloxicin

SUMMARY:
A Two-Part Phase 1 Study to Investigate A) Safety and Tolerability of Supratherapeutic dose of Zanubrutinib (BGB-3111) and B) Effect of Zanubrutinib on Cardiac Repolarization in Healthy Subjects

DETAILED DESCRIPTION:
This is a Two-Part Phase 1 Study.

Part A: This is a randomized, placebo-controlled, double blind, single dose study to evaluate the safety and tolerability of a single oral supratherapeutic dose of zanubrutinib in eight (8) subjects.

Part B: This is a randomized, placebo and positive-controlled, double-blind, 4-way crossover study being conducted in about 28 subjects to investigate the effect of a single therapeutic dose of zanubrutinib, a supratherapeutic dose of zanubrutinib and placebo on cardiac repolarization. Open-label Moxifloxacin (400 mg), a fluoroquinolone broad spectrum antibiotic will be used as a positive control.

ELIGIBILITY:
Inclusion Criteria: All subjects

1. Body mass index (BMI) 18 - 33 kg/m2, inclusive.
2. In good general health as assessed by the Investigator.
3. Females of non-child bearing potential.
4. Males without a vasectomy will agree to use required barrier contraception, and will agree to not donate sperm from the time of the first dose of BGB-3111 until ≥ 90 days after the last dose of BGB-3111.
5. Able to comprehend and willing to sign consent.

Exclusion Criteria: All subjects

1. Subjects with a clinically relevant history or presence of any clinically significant disease.
2. Personal or known family history of congenital or acquired long QT syndrome or cardiovascular disease.
3. Women of child-bearing potential.
4. History of alcoholism or drug/chemical abuse within 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of treatment-emergent adverse events (safety and tolerability) | Up to 8 days
  Incidence of treatment-emergent adverse events reported for zanubrutinib compared with placebo
Part B: Corrected QT interval [QTc] | Up to 2 days
  Evaluate the effects of single doses of zanubrutinib on the corrected QT interval [QTc] using the Fridericia correction [QTcF]) compared with placebo

SECONDARY OUTCOMES:
Part A: PK Parameters | Up to 3 days
  Plasma concentrations of zanubrutinib to evaluate protocol specified PK parameters
Part B: Heart Rate (HR) | Up to 2 days
  Evaluate the effects of a single dose of zanubrutinib and a single supratherapeutic dose of zanubrutinib on heart rate (HR)
Part B: PR Intervals | Up to 2 days
  Evaluate the effects of a single dose of zanubrutinib and a single supratherapeutic dose of zanubrutinib on PR
Part B: QRS Intervals | Up to 2 days
  Evaluate the effects of a single dose of zanubrutinib and a single supratherapeutic dose of zanubrutinib on QRS Intervals
Part B: PK Parameters | Up to 2 days
  Plasma concentrations of zanubrutinib to evaluate protocol specified PK parameters
Part B: Incidence of treatment-emergent adverse events (safety and tolerability) | Up to 16 days
  Incidence of treatment-emergent adverse events reported for zanubrutinib

CONTACTS AND LOCATIONS:
Overall Officials: William Novotny, MD, Study Director — BeiGene
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mu S, Darpo B, Tang Z, Novotny W, Tawashi M, Xue H, Willett M, Lin L, Sahasranaman S, Ou YC. No QTc Prolongation With Zanubrutinib: Results of Concentration-QTc Analysis From a Thorough QT Study in Healthy Subjects. Clin Transl Sci. 2020 Sep;13(5):923-931. doi: 10.1111/cts.12779. Epub 2020 Apr 8. PMID 32144955